CLINICAL TRIAL: NCT04251078
Title: Monitoring Mutational Burden in Low Risk MDS Patients Using Sequential Peripheral Blood Samples
Status: Recruiting | Type: Observational
Sponsor: Josep Carreras Leukaemia Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: N/A-NI-MDS-PI-13279
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Myelodysplastic Syndromes - Progression cohort: According to the literature (Greenberg et al, Blood. 2012), around 5-15% are expected to progress to high/very high-risk MDS subtype or to acute myeloid leukemia (AML). According to the total cohort of patients, it is expected that 20 of them would comprise this group and will be studied by targeted deep sequencing.
- Myelodysplastic Syndromes - Non Progression cohort: 20 patients without progression will be analyzed by targeted deep sequencing in order to find out if there are any differences in the mutational spectrum compared with those disease progression cases.

SUMMARY:
Myelodysplastic syndromes (MDS) are a heterogeneous group of clonal hematopoietic stem cell malignancies. Somatic cytogenetic and molecular aberrations and the evolution of subclonal malignant cell populations are responsible for the development and progression of MDS into acute myeloid leukemia.

Within only one decade the availability of new genome-wide technologies, like next generation sequencing (NGS), has revolutionized basic research. The routine clinical use of NGS analysis together with well-established diagnostic tools, like chromosome banding analysis or fluorescence in situ hybridization, will substantially add to existing diagnostic and prognostic criteria. This comprehensive combined approach could revolutionize the way we manage patient care. However, little is known about the application of such techniques in routine diagnostics and standards for such analyses are still missing.

In a recent publication from the research group, (Article DOI: 10.1002/ajh.25089) it was demonstrated that the analysis of peripheral blood cells (at diagnosis) by NGS is feasible and yields data that are equivalent to the results obtained from bone marrow cells (BMC), which is currently the gold standard for most molecular diagnostic analyses.

Not longer depending on the severe and for the patient painful collection of bone marrow aspirates now it is possible to perform comprehensive genetic analysis at short intervals on peripheral blood of MDS patients to detect and closely monitor patterns/pathways of clonal evolution of the malignant cell population in a routine diagnostic setting. It is expected that the obtained data from this study will substantially add to:

1. Understand the functional relevance of identified mutations and the implications of combined mutations.
2. Condense the findings from NGS together with data from established genetic methods (conventional cytogenetics, FISH) to a comprehensive view on MDS genetics and its dynamics considering strengths and weaknesses of each component of this approach.
3. Demonstrate that peripheral blood could be an appropriate sample to perform NGS follow-up studies.

In a series of very low, low and intermediate risk MDS patients from Spain it is intended to retrospectively perform NGS (targeted deep sequencing) of diagnosis and consecutive follow-up samples selecting those cases that showed signs of progression of the disease.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a heterogeneous group of clonal hematopoietic stem cell malignancies. Somatic cytogenetic and molecular aberrations and the evolution of subclonal malignant cell populations are responsible for the development and progression of MDS into acute myeloid leukemia.

Within only one decade the availability of new genome-wide technologies, like next generation sequencing (NGS), has revolutionized basic research. The routine clinical use of NGS analysis together with well-established diagnostic tools, like chromosome banding analysis or fluorescence in situ hybridization, will substantially add to existing diagnostic and prognostic criteria. This comprehensive combined approach could revolutionize patients management. However, little is known about the application of such techniques in routine diagnostics and standards for such analyses are still missing.

In a recent publication from the research group, (Article DOI: 10.1002/ajh.25089) it was demonstrated that the analysis of peripheral blood cells (at diagnosis) by NGS is feasible and yields data that are equivalent to the results obtained from bone marrow cells (BMC), which is currently the gold standard for most molecular diagnostic analyses.

Not longer depending on the severe and for the patient painful collection of bone marrow aspirates, now it is possible to perform comprehensive genetic analysis at short intervals on peripheral blood of MDS patients to detect and closely monitor patterns/pathways of clonal evolution of the malignant cell population in a routine diagnostic setting. It is expected that the obtained data from this study will substantially add to:

1. Understand the functional relevance of identified mutations and the implications of combined mutations.
2. Condense the findings from NGS together with data from established genetic methods (conventional cytogenetics, FISH) to a comprehensive view on MDS genetics and its dynamics considering strengths and weaknesses of each component of this approach.
3. Demonstrate that peripheral blood could be an appropriate sample to perform NGS follow-up studies.

In a series of very low, low and intermediate risk MDS patients from Spain it is intended to retrospectively perform NGS (targeted deep sequencing) of diagnosis and consecutive follow-up samples selecting those cases that showed signs of progression of the disease.

Methodology

Taking into account the incidence of MDS in the area, it is planned to collect samples from 100 MDS patients per year (during the first 2 years of the project) categorized as very low, low and intermediate risk.

All collected samples will be analyzed by conventional cytogenetics (routinely performed as part of the diagnostic tests) and also SF3B1 mutation analysis will be done in order to screen common alterations in low risk patients. In this way, a better characterization of the patients will be done and personalized treatment options according to each patient´s risk could be offered.

According to the literature, around 5-15% are expected to progress to high/very high-risk MDS subtype or to acute myeloid leukemia (AML). Only those cases that show signs of disease progression will be retrospectively analyzed by NGS.

The following criteria will be taken for patients enrollment:

Inclusion criteria:

* Patients categorized as very low, low or intermediate risk according to the Revised International Prognosis Scoring System for MDS (IPSS-R).
* Patients that meet the previous criteria and are not receiving any treatment or are receiving supportive care only (erythropoietin is accepted).

Exclusion criteria:

* Patients with "MDS with isolated del(5q)" diagnosis, according to 2017 World Health Organization Classification (WHO).
* Patients receiving any disease modifying therapies (e.g. hypomethylating agents).

Definition of progression: evolution to high/very high risk MDS subtype or to AML.

Peripheral blood (PB) and bone marrow (BM) samples will be collected and stored at the moment of diagnosis. PB samples will be collected every 6 months and at the time of progression of the disease (before receiving any treatment) BM sample will be also collected.

DNA extraction will be performed in diagnosis BM samples and SF3B1 gene will be analyzed by Sanger sequencing in all cases.

A total of 40 cases are estimated to be studied by NGS, 20 patients that are expected to show a progression of the disease and 20 patients without progression:

* Those cases that show progression of the disease will be retrospectively analyzed by NGS. Estimating that 10% of patients could progress, it is expected to include 10 new patients per year (during the two first years of the project) in the molecular analysis. This accounts a total of 20 patients after 2 years of follow-up.
* NGS will be performed in DNA from whole BM and PB paired samples at the moment of diagnosis and progression. Three PB follow-up samples in between will also be analyzed in order to track clonal dynamics. This accounts a total of 7 samples per each patient that progress (Figure 1).
* Additionally, 20 patients without progression will be analyzed in order to find out if there are any differences in the mutational spectrum compared with those disease progression cases. The same time points that were taken into account for those cases that progressed will be considered for these non-progression cases.

A panel of genes including disease relevant regions of the following 40 genes will be studied:

ASXL1, ASXL2, BCOR, BCORL1, BRAF, CALR, CBL, CEBPA, CSF3R, CSNK1A1, DNMT3A, EZH2, ETV6, FLT3, GATA1, GATA2, IDH1, IDH2, JAK2, KIT, KMT2A (MLL), KRAS, MPL, NF1, NPM1, NRAS, PTPN11, RAD21, RUNX1, SETBP1, SF3B1, SMC3, SRSF2, STAG1, STAG2, TET2, TP53, U2AF1,WT1, ZRSR2.

Patients and related samples data will be registered in a unique database. All clinical data will be collected according to the parameters defined by the Spanish Group of Myelodysplastic Syndromes (GESMD). All patients enrolled in the project will be requested to fill and sign an informed consent form for research purposes approved by the Ethical Committee of the ICO-Hospital Germans Trias i Pujol (Badalona, Barcelona, Spain). All protocols will be in accordance to the Declaration of Helsinki and the national normative of confidentiality of the data (LOPD).

The bioinformatic analyses will be performed at Josep Carreras Leukaemia Research Institute (IJC Campus ICO-GTIP. Badalona, Spain). Due to the amount of data, each analysis needs to be run in a cluster computing center, and stored in a special storage system which is follows the current laws for data protection in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients categorized as very low, low or intermediate risk according to the Revised International Prognosis Scoring System for MDS (IPSS-R).
* Patients that meet the previous criteria and are not receiving any treatment or are receiving supportive care only (erythropoietin is accepted).

Exclusion Criteria:

* Patients with "MDS with isolated del(5q)" diagnosis, according to 2017 World Health Organization Classification (WHO).
* Patients receiving any disease modifying therapies (e.g. hypomethylating agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taking into account the incidence of MDS in the area, it is planned to collect samples from 100 MDS patients per year (during the first 2 years of the project) categorized as very low, low and intermediate risk.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
SF3B1 status in the whole cohort (n=200) | 1 day
  SF3B1 gene will be analyzed by Sanger sequencing in all cases.
Targeted deep sequencing analysis of MDS low risk cases that showed progression of the disease (n=20) | 1 day
  Those cases that show progression of the disease will be retrospectively analyzed by NGS. Estimating that 10% of patients could progress, it is expected to include 10 new patients per year (during the two first years of the project) in the molecular analysis. This accounts a total of 20 patients after 2 years of follow-up.
  Targeted deep sequencing (panel of 40 myeloid related genes) will be performed in DNA from whole BM and PB paired samples at the moment of diagnosis and progression. Three PB follow-up samples in between will also be analyzed in order to track clonal dynamics. This accounts a total of 7 samples per each patient that progress.
Targeted deep sequencing analysis of MDS low risk cases that remained stable (no progression of the disease) (n=20) | 1 day
  20 patients without progression will be analyzed in order to find out if there are any differences in the mutational spectrum compared with those disease progression cases. The same time points that were taken into account for those cases that progressed will be considered for these non-progression cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Josep Carreras Leukaemia Research Institute, Badalona, Barcelona, Spain